CLINICAL TRIAL: NCT06178185
Title: Predicting Rapid Increases in Severity by Obligate Rotation & Improving Total Hip Expedited Elective Surgery (PRIORITEES); A Novel Study Evaluating Patients Awaiting Total Hip Arthroplasty
Brief Title: A Novel Study Evaluating Patients Awaiting Total Hip Arthroplasty (PRIORITEES)
Acronym: PRIORITEES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 868
Record Dates: First submitted 2023-06-29; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Hip Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hip replacements are one of the NHS's highest volume procedures, with ~14,000 operations per month before the onset of the COVID-19 pandemic. Delays to surgery can have significant implications; meaning increasing levels of pain and worsening quality of life.

As of January 2021, following the initial waves of the COVID-19 pandemic, 58,000 people had waited an average of 25 additional weeks for their total hip replacement.

The results of the study will hopefully help treating clinicians identify patients in whom there may be further deterioration if surgery is significantly delayed.

DETAILED DESCRIPTION:
Patients attending their routine pre-operative assessment clinic who meet the inclusion criteria will be invited to take part in the study by their direct clinical care team. If they provide their consent, they will first be examined for their maximum hip internal rotation possible when supine with hip and knee flexed at 90 degrees.

They will then be asked to sit in front of a camera placed at a height 2 to 3 feet (0.6 to 0.9 m) off the ground and stand 6 feet (1.8 m) away(6). Patients will be asked to spread their feet as far apart from each other whilst sitting straight with hips and knees at 90 degrees. A photograph will be taken of their neutral position, and another with their best attempt at internal rotation.

The internal rotation angle obtained along with the photo number will be documented on a data collection sheet with a hospital sticker, BMI, oxford hip score and EQ5D score completed that day.

At the end of the day, this information shall be collated & transcribed onto an excel spreadsheet for subsequent x-ray and photo review & measurement, anonymisation and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Native hip arthritis
* On the waiting list for elective total hip replacement surgery
* Able to give informed consent to participate
* Existing medical records demonstrating 2 AP Pelvic Xray images taken at least 3 months apart

Exclusion Criteria:

* Inability to consent to participation
* Previous surgical intervention on the joint in question.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients awaiting hip replacement surgery.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-06-27 (Estimated); Study Completion 2024-06-27 (Estimated)

PRIMARY OUTCOMES:
The primary aim of this study is to evaluate the factors, including obligate external rotation, that are associated with risk of progression in hip OA. | Participants attend clinic for a one-time clinic visit.
  The Deterioration Index (mm/week) will be calculated as the difference in average joint space width for the affected hip in AP X-Ray images taken at least 12 weeks apart, divided by the number of weeks between the X-Ray images assessed. The relationship with the parameters collated (age, BMI, KL grade, presence of OER) and DI will be evaluated to work out a cut-off value for high or low DI as part of the validation study.
  The DI will also be evaluated as regards a relationship to the OHS and EQ5D to assess if there is a correlation with metrics used to assess subjective outcome in this patient cohort.

SECONDARY OUTCOMES:
1-Develop a simple grading system based on the aforementioned results, to evaluate the feasibility of aiding clinicians in prioritising patients for THR. | For approximately for 1 year, through study completion.
  The secondary aims of the study will be evaluated by analysing the suitability of a grading system for risk of progression of hip OA, based on factors that lead to the highest DI values.
  The presence of OER will be evaluated and evidence of correlation to the photographic internal rotation angle, as well as quality of life scores will be assessed.
2-Validate the assessment of obligate external rotation remotely using a camera. | For approximately for 1 year, through study completion.
  Participants will first be examined for their maximum hip internal rotation possible when supine with hip and knee flexed at 90 degrees.
  They will then be asked to sit in front of a camera placed at a height 2 to 3 feet (0.6 to 0.9 m) off the ground and stand 6 feet (1.8 m) away(6). Patients will be asked to spread their feet as far apart from each other whilst sitting straight with hips and knees at 90 degrees. A photograph will be taken of their neutral position, and another with their best attempt at internal rotation.
  The internal rotation angle obtained along with the photo number will be documented on a data collection sheet with a hospital sticker, BMI, oxford hip score and EQ5D score completed that day.
  At the end of the day, this information shall be collated & transcribed onto an excel spreadsheet for subsequent x-ray and photo review & measurement, anonymisation and analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nikolova S, Harrison M, Sutton M. The Impact of Waiting Time on Health Gains from Surgery: Evidence from a National Patient-reported Outcome Dataset. Health Econ. 2016 Aug;25(8):955-68. doi: 10.1002/hec.3195. Epub 2015 May 26. PMID 26013773